CLINICAL TRIAL: NCT00002420
Title: A Phase II, 24-Week, Open-Label Study Designed to Evaluate the Pharmacokinetics, Safety, Tolerability, and Efficacy of Novel Combination Therapy With Videx (Didanosine), Zerit (Stavudine), Rescriptor (Delavirdine Mesylate), and MKC-442 (With or Without Hydroxyurea) for the Treatment of HIV-1- Infected Patients Who Failed Previous Protease Inhibitor Treatment
Brief Title: The Safety and Effectiveness of Didanosine Plus Stavudine Plus Delavirdine Mesylate Plus MKC-442 in HIV-Infected Patients Who Have Not Had Success With Protease Inhibitors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pharmacia and Upjohn (Industry); Triangle Pharmaceuticals (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 292E; ICC 603
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — emivirine; Hydroxyurea; Delavirdine; Stavudine; Didanosine

INTERVENTIONS:
Drug: Emivirine
Drug: Hydroxyurea
Drug: Delavirdine mesylate
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give MKC-442, didanosine (ddI), stavudine (d4T), and delavirdine (DLV) to HIV-positive patients.

DETAILED DESCRIPTION:
Patients receive a treatment regimen consisting of didanosine, stavudine, delavirdine, and MKC-442 for 24 weeks. During the study, patients are evaluated for changes from baseline in plasma HIV-1 RNA levels and lymphocyte subsets and for development of adverse events and toxicities. Samples for population pharmacokinetics are collected from all patients every 4 weeks. Patients who experience virologic failure may add hydroxyurea to their treatment regimen or be discontinued from the study. Patients who add hydroxyurea to their regimen and subsequently experience virologic failure are discontinued from the study. After Week 24, patients with documented virologic response are eligible to continue receiving study treatment until their plasma HIV-1 RNA levels return to baseline levels. For patients receiving hydroxyurea beginning at Week 24, visits are conducted at Weeks 28, 32, 36, and every 12 weeks thereafter. For patients who continue taking didanosine, stavudine, delavirdine, and MKC-442 or who have started hydroxyurea treatment between Weeks 12 and 20, follow-up visits are conducted every 12 weeks, or sooner if needed, until the patient permanently discontinues study treatment.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are at least 18 years old.
* Have experienced treatment failure on a previous anti-HIV drug combination that contained at least one protease inhibitor. Your viral load must be between 5,000 and 50,000 copies/ml after 6 months of continuous treatment with that drug combination.
* Agree to use a barrier method of birth control, such as condoms, during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of certain medical conditions, such as pancreatitis, peripheral neuropathy, seizure disorder, or AIDS-related cancer (except for Kaposi's sarcoma).
* Are allergic to any of the study drugs.
* Have ever taken certain anti-HIV medications including non-nucleoside reverse transcriptase inhibitors (NNRTIs), ddI, or d4T.
* Have taken certain other medications including interleukin-2, interferon or a vaccine within 30 days of study entry.
* Have received radiation therapy or chemotherapy within 30 days of study entry. (Local radiation therapy is allowed.)
* Abuse alcohol or drugs.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific Oaks Med Group, Beverly Hills, California, United States